CLINICAL TRIAL: NCT00521599
Title: A Study of the Therapeutic Equivalency of MF DPI 100 mcg and 200 mcg Inhalers in Corticosteroid-Dependent Subjects With Moderate Asthma
Brief Title: A Study of the Equivalent Effectiveness of 400 mcg Mometasone Furoate Using Two Different Dry Powder Inhalers in Moderate Asthmatics (Study P04828)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P04828
Record Dates: First submitted 2007-08-27; First posted 2007-08-28 (Estimated); Results first posted 2010-03-23 (Estimated); Last update posted 2024-05-23 (Actual); Status verified 2022-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Mometasone Furoate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- MF DPI 2 x 100 mcg BID (Experimental): 2 inhalations of mometasone furoate dry powder inhaler (MF DPI) 100 mcg plus 1 inhalation of placebo matching MF DPI 200 mcg twice daily (BID) for 8 weeks
  Interventions: Drug: Mometasone furoate dry powder inhaler; Drug: Placebo
- MF DPI 1 x 200 mcg BID (Experimental): 1 inhalation of mometasone furoate dry powder inhaler (MF DPI) 200 mcg plus 2 inhalations of placebo matching MF DPI 100 mcg twice daily (BID) for 8 weeks
  Interventions: Drug: Mometasone furoate dry powder inhaler; Drug: Placebo
- Placebo (Placebo Comparator): 2 inhalations of placebo matching mometasone furoate dry powder inhaler (MF DPI) 100 mcg plus 1 inhalation of placebo matching MF DPI 200 mcg twice daily (BID) for 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mometasone furoate dry powder inhaler
  Other Names: Asmanex
  Arms: MF DPI 1 x 200 mcg BID; MF DPI 2 x 100 mcg BID
Drug: Placebo

SUMMARY:
This study is a placebo-controlled study with 8-weeks of double-blind treatment of mometasone furoate dry powder inhaler (MF DPI) 200 mcg twice daily (BID) using two different inhalers, preceded by the Screening Period and by 2 weeks of open-label treatment with one inhalation of MF DPI 200 mcg twice daily in corticosteroid-dependent asthmatic subjects. The objective of this study is to evaluate the therapeutic equivalency of the 100 mcg and 200 mcg MF DPIs when providing the same total daily dose (400 mcg/day).

ELIGIBILITY:
Inclusion Criteria:

18 years of age, either sex, any race, with a diagnosis of asthma of at least 12 months' duration.

* Must be on a stable regimen of a medium daily dose of ICS for at least 4 weeks immediately prior to Screening. Medium daily doses of ICS are:

  * >500 to 1000 mcg beclomethasone CFC
  * >250 to 500 mcg beclomethasone HFA
  * >600 to 1000 mcg budesonide DPI
  * >1000 to 2000 mcg flunisolide
  * >250 to 500 mcg fluticasone
  * 400 mcg MF
  * >1000 to 2000 mcg triamcinolone acetonide.
* Must have a documented reversibility test obtained within 12 months prior to signing the informed consent form. Otherwise, to document a diagnosis of asthma and ensure the subject's responsiveness to bronchodilators, one of the following methods can be used at the Screening Visit, or thereafter, but prior to the Baseline Visit:

  * An increase in absolute FEV1 of >=12% and >=200 mL within 30 minutes of administration of 4 puffs of albuterol.
  * A PEF variability of >20%, expressed as a percent of the best and lowest morning pre-bronchodilator PEF over at least 1 week.
  * A diurnal variation in PEF of >20% based on the difference between the pre-bronchodilator AM value and the post-bronchodilator value from the evening before, expressed as a percentage of the mean daily PEF value any day during the Run-in Period.
* At Screening and Baseline, the subject's FEV1 must be >=60% predicted, when all restricted medications have been withheld for the appropriate intervals. If, based on the clinical judgment of the investigator, there is no harm in changing the subject's asthma therapy, subjects on LABAs must be willing to discontinue the LABA and be transferred to open-label treatment with MF MDI 200 mcg BID for 2 weeks prior to randomization.
* Clinical laboratory tests conducted at the Screening Visit must be within normal limits or clinically acceptable to the investigator/sponsor before the subject is instructed to start using open-label MF DPI run-in medication. A chest x-ray performed at the Screening Visit or any type of chest imaging within 12 months prior to the Screening Visit must be clinically acceptable to the investigator.
* A female of childbearing potential must be using a medically acceptable, adequate form of birth control. This includes: 1) hormonal contraceptives as prescribed by a physician (oral combined, hormonal implant); 2) medically prescribed IUD; 3) condom in combination with a spermicide (double-barrier method); 4) monogamous relationship with a male partner who has had a vasectomy. The subject must have started this birth control method at least 3 months prior to Screening (with the exception of condom in combination with spermicide), and must agree to continue its use for the duration of the study. A subject of childbearing potential who is not currently sexually active must agree and consent to using a medically acceptable method should she become sexually active during the course of this study. Women who have been surgically sterilized or are at least 1 year postmenopausal are not considered to be of childbearing potential. A subject of childbearing potential must have a negative serum pregnancy test at Screening.

Exclusion Criteria:

* A change in absolute FEV1 of >20% at any time from the Screening Visit up to and including the Baseline Visit.
* A clinical asthma exacerbation (defined as a deterioration of asthma that results in emergency treatment, hospitalization, or treatment with additional, excluded asthma medication at any time from the Screening Visit up to and including the Baseline Visit).
* Treatment in the emergency department or admission to the hospital for an asthma exacerbation 12 months prior to Screening.
* An upper or lower respiratory tract infection within the 4 weeks of to Screening. Visits can be rescheduled to meet this requirement.
* Evidence of clinically significant oropharyngeal candidiasis at Baseline with or without treatment. If there is evidence of oropharyngeal candidiasis at Screening and/or during the MF DPI Run-in Period, the subject may be treated as appropriate and the Baseline Visit can be scheduled upon resolution. If there is evidence of oropharyngeal candidiasis at the Baseline Visit, the subject may be treated as appropriate and the visit can be rescheduled upon resolution.
* A smoker or ex-smoker and has smoked within the previous year or has had a cumulative smoking history >10 pack-years.
* Requires more than twelve inhalations of albuterol or more than 2 treatments with nebulized beta-agonists on any 2 consecutive days during the Run-in Period.
* Ever required mechanical ventilation secondary to an asthma exacerbation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 672 (Actual)
Dates: Start 2007-05; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- MF DPI 1 x 200 mcg BID: 1 inhalation of MF DPI 200 mcg plus 2 inhalations of placebo matching MF DPI 100 mcg twice daily for 8 weeks
- Placebo BID: 2 inhalations of placebo matching MF DPI 100 mcg plus 1 inhalation of placebo matching MF DPI 200 mcg twice daily for 8 weeks
Period: Overall Study
Arm/Group | MF DPI 2 x 100 mcg BID | MF DPI 1 x 200 mcg BID | Placebo BID
Started | 268 | 268 | 136
Completed | 243 | 239 | 100
Not Completed | 25 | 29 | 36
Not completed — Adverse Event | 5 | 7 | 6
Not completed — Treatment Failure | 8 | 9 | 22
Not completed — Lost to Follow-up | 2 | 1 | 2
Not completed — Withdrawal by Subject | 3 | 5 | 1
Not completed — Withdrawal by subject treatment related | 3 | 1 | 2
Not completed — Protocol Violation | 2 | 4 | 2
Not completed — Did not meet protocol eligibility | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MF DPI 2 x 100 mcg BID | MF DPI 1 x 200 mcg BID | Placebo BID | Total
Number analyzed (Participants) | 268 | 268 | 136 | 672
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 259 | 255 | 131 | 645
  >=65 years | 9 | 13 | 5 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 182 | 178 | 104 | 464
  Male | 86 | 90 | 32 | 208

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Average AM Peak Expiratory Flow (PEF) Over the 7 Days of Week 8.
Description: Week 8 End = The last 7 days of data with the last day within the range of Days 51 to 64.
Time Frame: Baseline and Week 8 End
Population: All treated subjects included all but one placebo-treated subject from the All Randomized Subjects data set, who was randomized, but never treated in either the open-label or double-blind Treatment Periods due to non-compliance with the protocol
Measure: Least Squares Mean (Standard Deviation); unit: liters/minute
Arm/Group | MF DPI 2 x 100 mcg BID | MF DPI 1 x 200 mcg BID | Placebo BID
Number analyzed (Participants) | 268 | 268 | 136
liters/minute
  Baseline | 361.8 (96.7) | 374.3 (96.7) | 348.4 (96.7)
  Week 8 End | 6.03 (37.0) | 7.65 (37.0) | -7.93 (37.0)
Statistical Analysis 1: Comparison: MF DPI 2 x 100 mcg BID vs MF DPI 1 x 200 mcg BID; Week 8 End scores; Test type: Non-Inferiority or Equivalence — assume n=240 per group and standard deviation (STD) = 45 L/min for AM Peak Flow Rate at Week 8. If the two actives are the same, 95% CI of their mean difference has 90% probability to be completely within +/- 15 L/min; p = 0.654, ANOVA; Mean Difference (Net) = -1.62, 95% CI 2-sided [-8.74 to 5.49], Standard Deviation 37.0
Statistical Analysis 2: Comparison: MF DPI 2 x 100 mcg BID vs Placebo BID; Week 8 End scores; Test type: Superiority or Other; p = 0.003, ANOVA
Statistical Analysis 3: Comparison: MF DPI 1 x 200 mcg BID vs Placebo BID; Week 8 End scores; Test type: Superiority or Other; p = 0.001, ANOVA

ADVERSE EVENTS:
Groups:
- OL 1 X 200 mcg BID: Open-label MF DPI 200 mcg BID
- MF DPI 2 x 100 mcg BID: 2 inhalations of MF DPI 100 mcg plus 1 inhalation of placebo matching MF DPI 200 mcg twice daily for 8 weeks
- Placebo: 2 inhalations of placebo matching MF DPI 100 mcg plus 1 inhalation of placebo matching MF DPI 200 mcg twice daily for 8 weeks
Arm/Group | OL 1 X 200 mcg BID | MF DPI 2 x 100 mcg BID | MF DPI 1 x 200 Mcg BID | Placebo
Serious Adverse Events (participants affected / at risk) | 1/950 | 3/268 | 2/268 | 2/135
Other Adverse Events (participants affected / at risk) | 10/950 | 19/268 | 30/268 | 16/135
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OL 1 X 200 mcg BID (N=950) | MF DPI 2 x 100 mcg BID (N=268) | MF DPI 1 x 200 Mcg BID (N=268) | Placebo (N=135)
OESOPHAGEAL RUPTURE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CHEST PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
POST PROCEDURAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MULTIPLE INJURIES (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OPEN FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OL 1 X 200 mcg BID (N=950) | MF DPI 2 x 100 mcg BID (N=268) | MF DPI 1 x 200 Mcg BID (N=268) | Placebo (N=135)
NASOPHARYNGITIS (Infections and infestations) | 6 (6) | 10 (10) | 16 (16) | 6 (8)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 (4) | 10 (11) | 14 (14) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees not to publish or publicly present any interim results of the study without the prior written consent of sponsor. The investigator further agrees to provide the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication. The sponsor has the right to review and comment. If the parties disagree, the investigator agrees to meet with the sponsor's representative in order to resolve such issues.